CLINICAL TRIAL: NCT02645110
Title: Openly, Controlled Interventional Trial for Evaluating the Effectiveness of Whole-natural Hand-wash Formulations in Bacterial Removal and Openly Randomized Trial for Estimating the Relative Mildness of the Formulations
Brief Title: Evaluation of Effectiveness and Mildness of Whole-natural Hand-wash Formulations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mother's Choice Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0602-15-HMO
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Hand Hygiene; Skin Irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MC Hand soap (Experimental): For bacterial removal trial: Hand washing with the tested soap following bacterial application
  Interventions: Device: MC Hand Soap
- Water (Sham Comparator): For bacterial removal trial: Hand washing with tap water alone following bacterial application
  Interventions: Device: Tap water

INTERVENTIONS:
Device: MC Hand Soap — Washing hand with soap in comparison to hand washing with water alone
  Arms: MC Hand soap
Device: Tap water — Washing hand with water alone in comparison to hand washing with soap
  Arms: Water

SUMMARY:
The purpose of this study is to evaluate the effectiveness of whole-natural hand-wash formulations in bacterial removal and to estimate the relative mildness of the formulations.

DETAILED DESCRIPTION:
Hand washing with soap and water is one of the main ways to prevent the spread of diseases in general and specifically, the spread of hospital-acquired diseases. Mother's Choice Company develops natural products and technologies which include hand-wash soap. The purpose of this project is developing a whole-natural hand wash soap including no harmful ingredients which will succeed to remove at least 99.9% (3 log reduction) of the hand transient microbiota. In addition, the soap will be mild enough to allow the use of dozens times a day. The procedure for evaluating soap effectiveness in bacterial removal will include in general: bacterial application on hands, hand washing with the tested soap, sampling of hands before and after hand washing. The procedure for soap mildness estimation will include exposure of specific area of the arm or the back skin to the soap and following up and grading the reaction of the skin.

ELIGIBILITY:
Inclusion Criteria:

For effectiveness test:

* Healthy subjects aged 18-60 (both sexes).
* Subjects must have short natural nails.
* Subjects must remove all jewelry from their hands and forearms before participating.
* Subjects must not expose their hands to any antimicrobial products for 24 hours before the test (including antimicrobial containing dish soaps, shampoos, and body washes).
* Subjects must don safety glasses and lab coat prior to participating.
* Subjects will not be exposed to more than one challenge microorganisms per week and more than five challenge microorganisms in total.

For mildness test:

* Subject aged 18-60
* Subjects should be healthy adults from both sexes (preferably more women than men)
* Subjects would be able to participate in one study per four weeks.

Exclusion Criteria

For effectiveness test:

* Subjects cannot have any breaks or cuts in the skin of the hands or forearms.
* Subjects cannot have a medical diagnosis of a physical condition.
* Subjects cannot have allergies to detergents, hand hygiene products, perfume or any other substance they are going to be expose to.
* Subjects must not be on antibiotics or have been on antibiotics in the past 14 days.
* Subjects cannot participate if they have participated in other clinical trials within the past 14 days.
* Subjects cannot have any other general health or skin issues not mentioned above.
* Subjects cannot be pregnant or nursing.

For mildness test:

* pregnant or nursing subjects
* Subjects with an allergy or a skin disease which interferes with the proper results of the tests.
* Subjects who are taking medications which can interfere with the proper results of the tests. For example: systemic corticosteroids, topical steroids applied to the test area.
* Subjects with sun or phototherapy induced tanning at the test area.
* Subject who had been participating in allergy tests within four weeks prior to the present tests.
* Subjects could not use cosmetics for the face area except for the use of lipstick and makeup around the eyes for two weeks before the test.
* Subjects can use only mild soap and no more than once a day.
* Subjects should avoid drinking alcohol, coffee, tea and smoking on the test day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-03 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the tested hand-wash soaps in bacterial removal, presented as Log reduction | one year
  For log reduction determination the bacterial counts will be converted to log10. Next, the final quantity of bacteria recovered from hands after washing hands with the tested soap will be reduced from the start quantity of bacteria that was recovered from hands after bacterial application (before washing hands). For each soap the log reduction of each subject and the average log reduction will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Allon Moses, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Mother's Choice LTD, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes